CLINICAL TRIAL: NCT00078039
Title: Randomized, Double-blind, Placebo- and Active-controlled Parallel Group, Dose-response Study to Evaluate the Efficacy and Safety of 3 Fixed Dosages of Paliperidone Extended Release (6, 9, and 12 mg/Day) and Olanzapine (10 mg/Day) With Open-label Extension in Treatment of Schizophrenia
Brief Title: Trial Evaluating Three Fixed Dosages of Paliperidone Extended-Release (ER) Tablets and Olanzapine in the Treatment of Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003379
Record Dates: First submitted 2004-02-17; First posted 2004-03-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The primary objective of the double blind phase of this study is to evaluate the efficacy and safety of 3 fixed dosages of paliperidone ER (6, 9, and 12 mg/day) compared with placebo in adult patients with schizophrenia.

DETAILED DESCRIPTION:
Paliperidone is being developed as a new therapeutic agent for the treatment of schizophrenia. The ER formulation of paliperidone was developed to deliver paliperidone at a relatively constant rate over a 24-hour period to improve the tolerability profile and decrease the potential for orthostatic hypotension. This study is designed to evaluate the efficacy and safety of 3 fixed dosages of paliperidone ER (6, 9, and 12 mg/day) compared with placebo in patients with schizophrenia. This trial is a multicenter, double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), randomized (patients will be assigned to different treatment groups based solely on chance), placebo- and active-controlled, parallel-group, dose-response study. The study includes a screening period of up to 5 days, followed by double-blind treatment phase of 6 weeks. Following the double-blind treatment phase, eligible patients (those who have completed the 6-week double-blind phase or who discontinue due to lack of efficacy after a minimum of 21 days) may enter a 52-week open-label extension phase with paliperidone ER monotherapy. Patients will be randomly assigned to 1 of 5 treatments (paliperidone ER 6, 9, or 12 mg, olanzapine 10 mg, or placebo) and will take oral dosages of assigned treatment once daily during the 6-week double-blind period. At the time patients enter the double-blind period, they must be inpatients, and must remain in the hospital for a minimum of 14 full days. While patients are hospitalized, efficacy will be assessed twice during the first week and at the end of the second week. After patients are discharged from the hospital, they will return to have efficacy and safety assessments performed on a weekly basis through the end of the 6-week double-blind period. The efficacy response will be measured by the change in the PANSS total score from start of treatment to the end of the double-blind phase. Safety will be monitored throughout the study and includes assessments of the incidence of adverse events; measurement of extrapyramidal symptoms using 3 rating scales (Abnormal Involuntary Movement Scale [AIMS], Barnes Akathisia Rating Scale [BARS], Simpson-Angus Rating Scale [SAS]); measurement of vital signs (lying down and standing blood pressure, pulse, temperature); electrocardiograms; and clinical laboratory tests. Double-blind: 6-, 9-, or 12-mg fixed dose of paliperidone ER, olanzapine 10 mg or placebo taken orally once daily for 6 weeks.

Open-label extension: start on paliperidone ER 9 mg taken orally once a day; maintained on a flexible oral dosage of paliperidone ER (3, 6, 9, or 12 mg/day) for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Double-blind phase: DSM-IV diagnosis of schizophrenia at least 1 year prior to screening
* experiencing an acute episode, with a total PANSS score at screening between 70 and 120
* agree to voluntary hospitalization for a minimum of 14 days
* willing and able to fill out self-administered questionnaires
* able to be compliant with self-administration of medication, or have consistent help/support available.

Open-label extension phase: completed the 6 weeks of double-blind treatment or completed at least 21 days of treatment and discontinued due to lack of efficacy

* patient and investigator agree that open-label treatment is in the best interest of the patient.

Exclusion Criteria:

* Double-blind phase: DSM-IV axis I diagnosis other than schizophrenia
* DSM-IV diagnosis of substance dependence within 6 months prior to screening evaluation (nicotine and caffeine dependence are not exclusionary)
* history of tardive dyskinesia or neuroleptic malignant syndrome (NMS)
* history of any severe preexisting gastrointestinal narrowing (pathologic or iatrogenic)
* previous history of lack of response (2 adequate trials) to any antipsychotic
* significant risk of suicidal or violent behavior. Open-label phase: At significant risk for suicidal or violent behavior
* received an injection of a depot antipsychotic since entry into the preceding double-blind phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2004-03; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total PANSS score to the end of the double-blind phase.

SECONDARY OUTCOMES:
Assessment of global improvement in severity of illness; Evaluations of the benefits to quality of life; Assessment of the benefits to personal and social functioning. Incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Meltzer HY, Bobo WV, Nuamah IF, Lane R, Hough D, Kramer M, Eerdekens M. Efficacy and tolerability of oral paliperidone extended-release tablets in the treatment of acute schizophrenia: pooled data from three 6-week, placebo-controlled studies. J Clin Psychiatry. 2008 May;69(5):817-29. doi: 10.4088/jcp.v69n0515. PMID 18466043
- See also: Trial Evaluating Three Fixed Dosages of Paliperidone Extended-Release (ER) Tablets and Olanzapine in the Treatment of Patients With Schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=525&filename=CR003379_CSR.pdf